CLINICAL TRIAL: NCT05430243
Title: Empagliflozin in the Management of Cirrhosis-related Refractory Ascites: a Randomized Controlled Trial
Brief Title: Empagliflozin as a Novel Therapy in Refractory Ascites
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Kamal, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0305418
Record Dates: First submitted 2022-06-18; First posted 2022-06-24 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Ascites Hepatic
MeSH Terms: interventions — empagliflozin; Diuretics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empagliflozin group (Experimental)
  Interventions: Drug: Empagliflozin 10 MG; Drug: Diuretics
- standard treatment only group (Active Comparator)
  Interventions: Drug: Diuretics

INTERVENTIONS:
Drug: Empagliflozin 10 MG — once daily empagliflozin 10mg+/- diuretics
  Arms: Empagliflozin group
Drug: Diuretics — diuretics as clinically indicated

SUMMARY:
The aim of the present study is to investigate the safety, efficacy and cost-effectiveness of empagliflozin, a sodium glucose transporter 2 inhibitor, as an add on therapy to the standard care for refractory ascites in patients with liver cirrhosis

DETAILED DESCRIPTION:
Midodrine will be added if the blood pressure less than 100/70 mmHg during the follow up period (start by dose 5 mg three times daily and up titrate the dose according to the blood pressure monitoring to maximum dose 12.5 mg three times daily.

* Treatment of empagliflozin will be stopped if patient developed any of the following (attack of symptomatic hypoglycemia, hypotention not responding vasopresser agent, complicated urinary tract infection or attack of diabetic ketoascidosis) .
* The dose of diuretics will be reduced if marked weight reduction occurred (more than 0.5 kilogram/day in patient with ascites only or more than 1 killogram /day in patients with ascites and lower limb edema).
* The diuretics will be stopped temporally if any of the following (renal impairment, attack of hepatic encephalopathy, severe electrolyte imbalance) and permanently if the urine sodium < 30 mEq per day or there are intolerable side effects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age older than 18 years old. 2. Ability to give a written informed consent. 3. Decompensated liver cirrhosis complicated with ascites. 4. Diagnosis of refractory ascites has made 3 months before informed consent which defined as one of the following(6)

  1. Ascites that cannot be mobilized or the early recurrence of which cannot be prevented despite moderate salt restriction and maximum dose of diuretics ( furosemide 160 mg or equivalent and spironolactone 400mg)
  2. Ascites that cannot be mobilized or the early recurrence of which cannot be prevented because of the development of diuretic-induced complications that preclude the use of an effective diuretic dosage.

Exclusion Criteria:

* 1. History of any attack of hypoglycemia (defined as serum glucose less than 70 mg/dl) either symptomatic or a symptomatic.

  2. Blood pressure below 90/60 or History of Hypotension requiring high dose of vasopressor therapy (more than 15mg midodrine /day) 3. Patients who receive non-selective B-blockers. 4. History of recurrent urinary tract infection defined as more than 2 infections in last 6 months 5. Pregnancy and breast feeding 6. History of hypersensitivity to any SGLT2 inhibitor 7. Presence of hepatocellular carcinoma or any other malignancy. 8. eGFR below 30 ml/min using Modification of Diet in Renal Disease study (MDRD) 9. Patients with history of diabetes mellitus complicated with diabetic ketoacidois (DKA) or patients have any risk factors for DKA 10. History of alcohol intake 11. Modified Child-Pugh score 12 or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
No need for paracentecis | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt